CLINICAL TRIAL: NCT02855138
Title: The Effects of Oral Isotretinoin in Women With Acne and Polycystic Ovary Syndrome
Brief Title: Effects of Isotretinoin on The Gonads and Hirsutism
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kayseri Education and Research Hospital (Other Government)
Collaborators: Kayseri Erciyes University Faculty of Medicine (Unknown)
Responsible Party: Principal Investigator, Gökhan Açmaz, obstetrics and gynecology, Kayseri Education and Research Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2016/358
Record Dates: First submitted 2016-08-01; First posted 2016-08-04 (Estimated); Last update posted 2016-08-05 (Estimated); Status verified 2016-07

CONDITIONS: Adverse Effects of Medical Drugs
Keywords: isotretinoin; PCOS; acne vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Isotretinoin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor

ARMS (2):
- study group (Active Comparator): The study group consisted of 40 volunteers women with PCOS (aged 18- 40 years, BMI, 18-44kg/m2) who attended the obstetrics and gynecology clinic for the treatment of menstrual irregularities and hirsutism.The patients were treated with 0.6-0.8 mg/kg oral isotretinoin up to a total dose of 120-150 mg/kg. Treatment was started at 20 mg/day and gradually increased to the maximum of 40 mg/day. The patients were monitored monthly during isotretinoin treatment.
  Interventions: Drug: oral isotretinoin
- control group (No Intervention): The control group of this study was pretreatment period of the same volunteer patients.

INTERVENTIONS:
Drug: oral isotretinoin
  Other Names: roaccutane
  Arms: study group

SUMMARY:
The investigators consider that there are some rising concerns about the use of isotretinoin by women of reproductive age with depleted ovarian reserve, hence it is important to detect the effect of isotretinoin on ovarian reserve.

There has not been a well-designed study evaluating its effects on the human ovarian reserve, hormone levels and menstrual cycles in women with polycystic ovary syndrome (PCOS). For this reasons, this study was administered to determine whether there is an effect of isotretinoin on the gonads and hirsutism in women with acne and PCOS.

ELIGIBILITY:
Inclusion Criteria:

* consisted of 40 volunteers women with PCOS (aged 18- 40 years, BMI, 18-44kg/m2) who attended our obstetrics and gynecology clinic for the treatment menstrual irregularities and hirsutism

Exclusion Criteria:

* 1)presence of any dermatologic disorder besides acne 2) presence of any systemic disease 3) exposure to any systemic treatment in the last three months that could alter ovarian reserve 4) pregnancy or lactation 5) infection diseases 6) use of antidepressants, steroidal hormone drugs, mood stabilizers, caffeine, alcohol, or tobacco 7) histories of abdominal surgery for endometriosis or ovarian surgery

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2015-01; Primary Completion 2016-03 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Adverse Events on the Gonads and Hirsutism That are Related to Treatment | six months

CONTACTS AND LOCATIONS:
Overall Officials: GÖKHAN ACMAZ, Principal Investigator — Kayseri Education and Research Hospital

REFERENCES:
- [Derived] Acmaz G, Cinar L, Acmaz B, Aksoy H, Kafadar YT, Madendag Y, Ozdemir F, Sahin E, Muderris I. The Effects of Oral Isotretinoin in Women with Acne and Polycystic Ovary Syndrome. Biomed Res Int. 2019 Apr 7;2019:2513067. doi: 10.1155/2019/2513067. eCollection 2019. PMID 31080813